CLINICAL TRIAL: NCT02355015
Title: A Prospective Registry For Non Tuberculous Mycobacterial (NTM) Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/205/F
Record Dates: First submitted 2015-01-28; First posted 2015-02-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Mycobacterium Infections, Nontuberculous
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to address the following aims

1. To provide an overview of the epidemiology of the patients who are managed in the Singapore General Hospital for NTM infections.
2. To evaluate the medical care of patients in the institution with regards to the type of medical and/or surgical treatment received and specifically, the antibiotic regime and duration administered.
3. A longitudinal follow up which will allow an assessment of our care and patient outcome in this population cohort

DETAILED DESCRIPTION:
Nontuberculous Mycobacteria (NTM) is difficult to treat and has no standardised antibiotic therapy. There have been increasing recognition of the need for measurements of NTM care around the world, as rates of NTM infections have begun to supercede Tuberculosis infections for the first time. As health care-associated NTM outbreaks also pose an infection control risk for patients undergoing surgery, this study provides a platform for further greater uniformity and opportunities for improvement in care. (1,2)

Singapore General Hospital (SGH) is a tertiary hospital and sees patients of various complex medical illnesses. Patients with Nontuberculous Mycobacteria (NTM) infections are also on follow up with the infectious diseases specialists SGH. The care of NTM patients can last many years, with patients requiring multiple admissions for reinfections/relapses and are often on long term suppressive therapy and follow up at the Specialist Outpatient Clinic. (3,4)The lack of standardised care for NTM patients, lengthy treatment time for NTM infections, as well as increases in macrolide-resistant NTM infections, warrants a need for research into the epidemiology and best practice to treat this group of patients. (5,6) We seek to better define the epidemiology of this group of patients and hope to objectively measure the effectiveness and quality of our NTM care delivery in SGH.

Currently there is a lack of a systematic database to track our quality of care and support services. As there are many Infectious Diseases Specialists in the department, each may have slight variation in clinical practice and preference in the face of a lack of proper treatment guideline. We believe NTM management can be improved with a consistent care delivery pathway and more standardization of therapy and follow up plan. This will lead to better desired patient outcome. This prospective observational data collection will allow us to evaluate our current standard of care for these patients, which can lead to identification for areas of improvement so that we can refine our strategies and implement more effective and standardized guidelines in the future.

1. Griffith DE, Aksamit T, Brown-Elliott BA, Catanzaro A, Daley C, Gordin F, Holland SM, Horsburgh R, Huitt G, Iademarco MF, Iseman M, Olivier K, Ruoss S, von Reyn CF, Wallace RJ Jr, Winthrop K. An Official ATS/IDSA Statement: Diagnosis, Treatment, and Prevention of Nontuberculous Mycobacterial Diseases. Am J Respir Crit Care Med 2007; Feb 15;175(4):367-416
2. Cook JL. Nontuberculous mycobacteria: opportunistic environmental pathogens for predisposed hosts. Br Med Bull 2010;96:45-59
3. Piersimoni C. Nontuberculous mycobacteria infection in solid organ transplant recipients. European Journal of Clinical Microbiology & Infectious Diseases 2012 Apr;31(4):397-403
4. Payen MC, De Wit S, Clumeck N. Manifestations, diagnosis and treatment of non-tuberculous mycobacterial infections in patients with HIV infection. Revue des Maladies Respiratoires 1997 Dec;14 Suppl 5:S142-51
5. Russell CD, Claxton P, Doig C, Seagar AL, Rayner A, Laurenson IF. Non-tuberculous mycobacteria: a retrospective review of Scottish isolates from 2000 to 2010. Thorax 2013 [Epub ahead of print]
6. Binder AM, Adjemian J, Olivier KN, Prevots DR. Epidemiology of Nontuberculous Mycobacterial Infections and Associated Chronic Macrolide Use among Persons with Cystic Fibrosis. American Journal of Respiratory and Critical Care Medicine 2013; [Epub ahead of print]

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with Nontuberculous Mycobacteria infections.

Exclusion Criteria:

* Patient refusal to participate in the study

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with NTM infection in the institution
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 5 years
  Patients will be followed up on an outpatient basis and mortality outcomes (all cause) at 6 months, 1 year and 5 years will be monitored.

SECONDARY OUTCOMES:
Clinical response | 6 months from start of treatment
  Managing clinician will judge the clinical response post-induction and post-maintenance treatment. Responses classified as resolved, improved, stable or worse.
Microbiological response | 6 months from start of treatment
  This is specifically for NTM infections involving the lung. Sputum samples will be collected regularly in the 6 month period to document clearance of NTM growth from the sputum. A microbiological response would be classified as 2-3 negative consecutive sputum cultures in the 6 month period.
Chest Xray changes | 6 months
  This is specifically for NTM infections involving the lung. Chest Xray post completion of treatment will be assess and classified as resolved, improved, stable or worse.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Dr Cherng, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore